CLINICAL TRIAL: NCT06220318
Title: A Phase I/II Clinical Study on the Safety, Tolerability and Preliminary Efficacy of C019199 in Combination With Sintilimab in Patients With Advanced Solid Tumors
Brief Title: Assessment of the Safety and Efficacy of C019199 Plus Sintilimab in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujian Haixi Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXP019-CTPI-02
Record Dates: First submitted 2024-01-14; First posted 2024-01-23 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: DRUG: C019199
  The C019199 will be taken orally, once a day
  DRUG: Sintilimab
  Sintilimab will be administrated with intravenous infusion, 200mg, every 3 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C019199 plus Sintilimab (Experimental): Patients with selected tumors will received oral C019199 at a starting dose of 100mg once daily in combination with intravenous Sintilimab 200mg every 3 weeks ( Q3W ) on a 21-day treatment cycle until disease progression, development of unacceptable toxicity, or withdrawal of consent .
  Interventions: Drug: C019199; Drug: Sintilimab

INTERVENTIONS:
Drug: C019199 — The C019199 will be taken orally, once a day
  Other Names: C019199 Tablets
Drug: Sintilimab — Sintilimab will be administrated with intravenous infusion, 200mg, every 3 weeks.
  Other Names: IBI308

SUMMARY:
This is a phase I/II non-randomized, open-label, single-arm, multicenter study to evaluate the Safety and Efficacy of C019199 Plus Sintilimab in Participants With Advanced Solid Tumors.

DETAILED DESCRIPTION:
Phase I will determine and confirm the maximum tolerated dose(MTD) and recommended phase II dose(RP2D) for C019199 in combination with 200 milligrams (mg) ( intravenous[IV], every 3 weeks [Q3W]) Sintilimab in patients with advanced Solid tumors.

Phase II will evaluate the safety and efficacy of the combination of C019199 and Sintilimab in selected solid tumors at the RP2D from Phase I.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Age ≥18 years and <76 years at the time of signing informed consent, male or female;
2. Histologically or cytologically confirmed locally advanced or metastatic solid tumors that have progressed on or intolerant to standard therapy or whom no standard therapy exists;
3. ECOG score: 0-1;
4. Life expectancy of 3 months or more;
5. Phase II: have measurable disease based on RECIST 1.1 ;
6. Phase II: agree to provide archival tumor tissue or newly obtained biopsy of a tumor lesion ;
7. Have adequate organ function ;
8. A male or female participant must agree to use contraception during the treatment period and for at least 6 months after the last dose of study treatment ;
9. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

Subjects meeting any of the following criteria must be excluded from this study:

1. Known hypersensitivity to CSF-1R inhibitors or Sintilimab;
2. Receipt of (or planned receipt of) anti-tumor therapies within 4 weeks prior to first dose through the end of the study treatment period;
3. Incomplete recovery from prior therapy toxicities (i.e. grade 2 or higher toxicities at screening, except for alopecia, pigmentation changes, or immune-mediated hypothyroidism that is stable with hormone replacement);
4. History of malignancies other than the cancer being treated in this study (Exceptions include: malignancies that have been cured with no recurrence within 3 years prior to enrollment; completely resected basal cell or squamous cell skin cancer; any completely resected carcinoma in situ);
5. Major surgery (grade III or IV surgery) within 4 weeks prior to first dose without complete recovery;
6. History of prior surgeries or severe gastrointestinal diseases such as dysphagia, active gastric ulcers, ulcerative colitis, Crohn's disease, intestinal obstruction etc., that may affect absorption, distribution, metabolism of study treatment per investigator's judgement;
7. Any significant clinical or laboratory abnormalities that are considered clinically significant per investigator's judgement and make the subject unsuitable for enrollment, such as: uncontrolled active infections (CTCAE v5.0 grade 2), uncontrolled diabetes (fasting blood glucose >7.8 mmol/L despite optimal medical therapy), uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg despite optimal medical therapy), peripheral neuropathy ≥ grade 2 (CTCAE v5.0), congestive heart failure ≥ grade 2 (CTCAE v5.0), myocardial infarction within the last 6 months, severe/unstable angina or coronary/peripheral artery bypass graft, arterial thromboembolism or deep vein thrombosis, stroke and/or transient ischemic attack, moderate to severe hepatic cirrhosis, uncontrolled major seizure disorders, known history of autoimmune disease that is active or may relapse (except for clinically stable hypothyroidism);
8. Known active infection of human immunodeficiency virus (HIV) or hepatitis C virus (HCV);
9. For hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive subjects, HBV DNA level above upper limit of reference range;
10. Pregnant or lactating women;
11. Severe psychological or psychiatric abnormalities that may affect compliance with study requirements;
12. Detection of active or untreated CNS metastases on baseline imaging assessments by CT or MRI during screening: a) If new asymptomatic CNS metastases are detected on baseline scans, subjects must receive radiotherapy and/or surgery for CNS metastases, and can be enrolled without repeat CNS imaging if meeting all other criteria; b) Subjects with history of treated brain or meningeal metastases can be enrolled if clinically stable for at least 2 months and systemic high-dose corticosteroids (>10 mg/day prednisone or equivalent) has been discontinued for at least 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Cycle 1 (Cycle length=21 days)
  Dose-limiting toxicity (DLT) refers to a drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose.
Objective Response Rate (ORR) Based on iRECIST | From date of enrollment until the date of first documented progression or death
  ORR was defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) for target and non-target lesions.
Progression-free Survival (PFS) after administration | From date of enrollment until the date of first documented progression or death
  Progression-free Survival (PFS) is defined as the time from the date of first dose of the study drug to the first documented disease progression (according to iRECIST ) or death (due to any cause), whichever occurs first.

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events( TEAEs )and Serious Adverse Events （SAEs） | From the first dose until 28 days after the last dose
  A TEAE was defined as an adverse event (AE) that emerged during the time from the first dose of study drug to 28 days following the last dose of study drug,which does not necessarily have a causal relationship with the treatment. A Serious AE is any untoward medical occurrence that at any dose: resulted in death; was life threatening (that is, the participant was at immediate risk of death from the AE as it occurred; this does not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death) required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or is medically important due to other reasons than the above mentioned criteria
Cmax | Cycle 1 Day 1; Cycle 1 Day 21
  Maximum Plasma Concentration
AUC(0-t): | Cycle 1 Day 1; Cycle 1 Day 21
  Area under the concentration-time curve (AUC)
T1/2 | Cycle 1 Day 1; Cycle 1 Day 21
  Terminal Half-life
Disease Control Rate (DCR) after administration | From date of enrollment until the date of first documented progression or death
  Disease Control Rate (DCR) is defined as the proportion of patients with complete response, partial response and stable disease.
Duration of Remission (DoR) after administration | From date of enrollment until the date of first documented progression or death
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (PR or better) to the first documented disease progression evidence (according to iRECIST ) of the responders (who achieve PR or better response).se).
Overall Survival (OS) after administration | The time from the date of enrollment until death
  OS is defined as the time from the date of study treatment to the date of death due to any cause .

CONTACTS AND LOCATIONS:
Overall Officials: FENG YE, Principal Investigator — The First Affiliated Hospital of Xiamen University; YONGCHANG ZHANG, Principal Investigator — Hunan Cancer Hospital
Locations (2):
- China (2):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No